CLINICAL TRIAL: NCT03345212
Title: Implementation and Effect of Exercise and Respiratory Training on 6-minute Walking Distance in Patients With Severe Chronic Pulmonary Hypertension: a Randomized Controlled Multicenter Trial in European Countries
Brief Title: A Randomized Controlled Multicenter Trial of Exercise Training in Pulmonary Hypertension in European Countries
Acronym: EU-TRAIN-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EU-TRAIN-01
Record Dates: First submitted 2017-07-27; First posted 2017-11-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients in this group continue their sedentary life-style throughout the study period. Patients will be advised to perform no specific exercise training during the trial. After 15 weeks, the patients are offered to take part in the training program as well.
- Training group (Experimental): Standard rehabilitation therapy includes dietary measures, massages and relaxation techniques. Additionally, patients perform exercise and respiratory therapy and mental gait training.
  Patients will be informed about group allocation.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — The rehabilitation program comprises interval ergometer training, dumbbell training, respiratory therapy, mental training and guided walks for 5-7 times/week.
  Arms: Training group

SUMMARY:
Chronic pulmonary hypertension (PH) is associated with impaired exercise capacity, quality of life and right ventricular function. The disease is characterized by an increase of pulmonary vascular resistance and pulmonary arterial pressure, leading to right heart insufficiency.

Despite optimized combination-medical therapy most patients remain symptomatic, have reduced exercise capacity, quality of life and reduced survival rates, with an annual mortality rate of approximately 5 -15 % or even higher.

Previous training studies have suggested that exercise training as add-on to medical treatment is highly effective improving exercise capacity, quality of life and symptoms.

The current guidelines recommend exercise training only in specialized centres including both PH and rehabilitation specialists who are experienced in exercise training of severely compromised patients.

A specialized PH-training program has been performed in Heidelberg since 2003 including >1200 patients with various forms of chronic PH. The exercise training program is performed in a special setting with an in-hospital start of the rehabilitation program. It is characterized by a low-dose closely supervised exercise training in small groups with additional psychological support and mental training.

This training program for patients with PH will be implemented in European centers to add exercise training to the existing PH therapies. The effect of the training on physical exercise capacity will be assessed by 6-minute walking distance (6-MWD). Further clinical parameters will be assessed to evaluate the effect on exercise capacity, quality of life and symptoms.

The aim of this study is to guide European PH-centers to become specialized centers for training in PH.

126 patients will be included, who either receive exercise training or continue their daily sedentary life style (1:1 randomization) for 15 weeks.

As inpatient settings are not available in all healthcare systems the training program will be adapted from the specific training program for PH patients developed in Heidelberg to a procedure, which is feasible in the local participating centres. Another objective of this study is to assess if the particular adopted training program specified for each participating centre and country is still safe and effective.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is defined as a mean pulmonary arterial pressure ≥25 mmHg. PH is often diagnosed at an advanced stage (WHO functional class III-IV) with a massive increase of the mean pulmonary arterial pressure. A crucial parameter determining the symptoms and prognosis of the patients is the cardiac reserve. This parameter is defined by the pulmonary vascular resistance and the right ventricular adaptation. Severe PH is characterized by a decreased cardiac output at rest, an increased afterload and consecutive cor pulmonale.

Within the last years there has been a huge progress in the scientific fields of genetics, pathogenesis, pathophysiology and therapy of PH. This has also been documented in the PH world conferences. New disease-targeted medication has been developed such as endothelin receptor antagonists (bosentan, ambrisentan, sitaxentan, macitentan), prostacyclin derivates (inhaled and intravenous iloprost, epoprostenol, treprostinil), phosphodiesterase-5-inhibitors (sildenafil, tadalafil) and the soluble guanylate cyclase inhibitor riociguat. Despite these advances in treatment, the disease may not be treated causally or even be cured. In most cases however, disease progression may be slowed down. The use of PH-targeted treatment and supporting therapies such as anticoagulation and diuretics improve the symptoms and impede the progression of the disease. Nevertheless, the prognosis of the patients remains impaired. The first randomized controlled study investigating the effect of exercise training in PH showed a significant improvement of exercise capacity and quality of life. Further uncontrolled trials using a low-dose exercise and respiratory therapy in different etiologies of PH showed an improvement in exercise capacity, quality of life, muscle function and further prognostic parameters. A recent randomized controlled study could support these findings. Studies also showed an improvement in muscle capillarization of the quadriceps muscle.

The training program consists of interval ergometer training, respiratory therapy, muscle training and mental gait training. The interval ergometer training allows performing aerobic exercise training with a low cardio-circulatory stress. In patients with left heart insufficiency, this training has been successfully implemented. Respiratory therapy has been established in the rehabilitation of patients with lung disease within the last years. The different techniques aim to improve ventilation, strengthen the respiratory muscles, mobilize the thorax and enhance secretolysis. The training program also contains mental (gait) training. This training was adapted from mental imagery techniques used by sport psychologists in professional athletes. Mental imagery techniques have shown to improve physical and cognitive functions.

Due to the beneficial results, exercise training and rehabilitation has received a 1A recommendation at the PH world symposium in Nice in 2013. This decision was mainly based on three randomized controlled trials that investigated a limited number of patients. To unequivocally demonstrate safety and positive effects of exercise training in different settings large multicenter RCTs are essential. An exercise program has not yet been implemented in most European countries, partly due to limited access to rehabilitation programs and institutions.

The aim of this large, multicenter, prospective, randomized controlled trial is to investigate the effect of exercise training and rehabilitation on physical exercise capacity across different European countries. Physical exercise capacity will be measured by exercise induced change of 6-minute walking distance (6-MWD) compared to baseline and the control group without training. As inpatient settings are not available in all healthcare systems the training program will be adapted from the specific training program for PH patients developed in Heidelberg in a system, which is feasible for the local participating centres. Another objective of this study is to assess if the adopted training program specified for each participating centre and country is still safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients of any ethnic origin ≥ 18 years
* WHO functional class II-IV
* PH diagnosed by right heart catheter showing:

  * Baseline mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
  * Baseline pulmonary vascular resistance (PVR) ≥ 240 dyn x s x cm-5
  * Baseline pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg
* Patients receiving optimized conventional PH therapy including intensified treatment with diuretics and who have been stable for 2 months before entering the study
* Except for diuretics, medical treatment should not be expected to change during the entire 15-week study period
* Negative pregnancy test (β-HCG) at the start of the trial and appropriate contraception throughout the study for women with child-bearing potential
* Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria:

* PH of any cause other than permitted in the entry criteria, e.g. concomitantly to portal hypertension, complex congenital heart disease, reversed shunt, HIV infection, suspected pulmonary veno-occlusive disease based on pulmonary edema during a previous vasoreactivity test or on abnormal findings compatible with that diagnosis (septal lines or pulmonary edema at high resolution computer tomography), congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension or unclear diagnosis
* Pregnancy
* Patients with signs of right heart decompensation
* Walking disability
* Acute infection
* Pyrexia
* Any change in disease-targeted therapy within the last 2 months
* Any subject who is scheduled to receive an investigational drug during the course of this study
* Severe lung disease: FEV1/FVC <0.5 and total lung capacity < 70% of the normal value
* Active liver disease, porphyria or elevations of serum transaminases >3 x ULN (upper limit of normal) or bilirubin > 1.5 x ULN
* Hemoglobin concentration of less than 75 % of the lower limit of normal
* Systolic blood pressure < 85 mmHg
* Active myocarditis, instable angina pectoris, exercise induced ventricular arrhythmias, decompensated heart failure, hypertrophic obstructive cardiomyopathy, highly impaired left ventricular function
* History or suspicion of inability to cooperate adequately. will be excluded from the study.

Additional exclusion criteria for MRI (optional)

* Acute psychosis or other states of mind, which seem to impair patient's ability to comprehend instructions
* Patients with metal cardiac valves or other metal implants, incorporated ferromagnetic materials or MRI-incompatible active medicinal products
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
6 MWD | 15 weeks
  Change in 6-MWD between baseline and 15 weeks in the training vs. the control Group; meters

SECONDARY OUTCOMES:
Change in WHO functional class in training vs. control group | 15 weeks
  WHO functional class
Change in Quality of life in training vs. control group | 15 weeks
  Quality of life (SF-36)
Change in Borg scale 6-MWD training vs. control group | 15 weeks
  Borg scale 6-MWD
Change in tricuspid annular plane systolic excursion | 15 weeks
  Echocardiographic parameter training vs. control Group; mm
Change in tissue Doppler imaging | 15 weeks
  Echocardiographic Parameter training vs. control group
Change in left ventricular pump function | 15 weeks
  Echocardiographic Parameter training vs. control Group; qualitative
Change in right ventricular pump function | 15 weeks
  Echocardiographic Parameter training vs. control Group; qualitative
Change in thickness of interventricular septum | 15 weeks
  Echocardiographic Parameter training vs. control Group; mm
Change insize of inferior vena cava | 15 weeks
  Echocardiographic Parameter training vs. control Group; mm
Change in systolic pulmonary arterial pressure | 15 weeks
  Echocardiographic Parameter training vs. control Group; mmHg
Change in left ventricular eccentricity index | 15 weeks
  Echocardiographic Parameter training vs. control group
Change in Tei index | 15 weeks
  Echocardiographic Parameter training vs. control group
Change in right ventricular area | 15 weeks
  Echocardiographic Parameter training vs. control group
Change in right atrial area | 15 weeks
  Echocardiographic Parameter training vs. control Group; square cm
Change in workload | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry) training vs. control Group; Watts
Change in heart rate | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry) training vs. control Group; bpm
Change in ventilation | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry) training vs. control Group; L/min
Change in carbon dioxide output | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry) training vs. control Group
Change in spiroergometry parameters in training vs. control group | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry): VO2 at anaerobic threshold determined by V-slope method
Change in VCO2 at anaerobic threshold | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry): determined by V-slope method
Change in oxygen uptake | 15 weeks
  Cardiopulmonary exercise testing (spiroergometry); L/min/kg
Change in diffusion-limited carbon monoxide (DLCO) | 15 weeks
  Lung function; Diffusion capacity
Change in alveolar volume (VA) | 15 weeks
  Lung function
Change in residual volume (RV) | 15 weeks
  Lung function
Change in total lung volume (TLC) | 15 weeks
  Lung function
Change in forced expiratory flow | 15 weeks
  Lung function
Change in peak expiratory flow rate | 15 weeks
  Lung function
Change in forced expiratory volume in one second (FEV1) | 15 weeks
  Lung function; total and in percentage
Change in forced vital capacity (FVC) | 15 weeks
  Lung function
Change in NTproBNP | 15 weeks
  Laboratory marker for the impairment of the right heart
Change in interleukins | 15 weeks
  Laboratory marker for the impairment of the right heart
Change in inflammatory markers | 15 weeks
  Laboratory marker for the impairment of the right heart
Change in carbon dioxide partial pressure | 15 weeks
  Blood gas Analysis
Change in oxygen saturation of the blood (SaO2) | 15 weeks
  Blood gas analysis
Change in additional oxygen supplementation (yes/no and quantity) | 15 weeks
  Blood gas analysis
Change in oxygen partial pressure | 15 weeks
  Blood gas analysis
Change in oxygen saturation | 15 weeks
  Safety Parameter; L/min
Assessment of clinical laboratory Investigation alerts (values out of range) | 15 weeks
  Safety parameter
Assessment of adverse Events | 15 weeks
  Safety Parameter; unrelated and related to procedure
Assessment of serious adverse events | 15 weeks
  Safety parameter
frequency of hospitalizations | 15 weeks
  Safety parameter
length of hospitalizations | 15 weeks
  Safety parameter
Change in resting heart rate | 15 weeks
  Safety parameter
Change in blood pressure | 15 weeks
  Safety parameter
frequency of pathological findings in long-term ECG | 15 weeks
  Safety parameter
Qualitative Review of electrocardiogram (ECG) | 15 weeks
  Safety Parameter; pathological findings
Assessment of survival | 1 year
  Training and control Group; transplant-free and Overall survival
Change of the right ventricular size | 15 weeks
  Optional: Changes in MRI parameters
Change of the right ventricular pump function | 15 weeks
  Optional: Changes in MRI parameters
Change of the left ventricular size | 15 weeks
  Optional: Changes in MRI parameters
Change of the left ventricular pump function | 15 weeks
  Optional: Changes in MRI parameters
Change in microRNA expression | 15 weeks
  Optional: Epigenetic changes
Change in DNA-methylation | 15 weeks
  Optional: Epigenetic changes
Assessment of relationship of DNA mutations and disease progression | 15 weeks
  Optional: Investigation of DNA mutations relationship to disease progression
Assessment of relationship of DNA mutations and training effects | 15 weeks
  Optional: Investigation of DNA mutations

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, MD, Principal Investigator — Centre for pulmonary hypertension of the Thoraxclinic at the University Hospital Heidelberg
Locations (1):
- Centre for pulmonary hypertension of the Thoraxclinic at the University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Background] Grunig E, Ehlken N, Ghofrani A, Staehler G, Meyer FJ, Juenger J, Opitz CF, Klose H, Wilkens H, Rosenkranz S, Olschewski H, Halank M. Effect of exercise and respiratory training on clinical progression and survival in patients with severe chronic pulmonary hypertension. Respiration. 2011;81(5):394-401. doi: 10.1159/000322475. Epub 2011 Feb 9. PMID 21311162
- [Background] Grunig E, Lichtblau M, Ehlken N, Ghofrani HA, Reichenberger F, Staehler G, Halank M, Fischer C, Seyfarth HJ, Klose H, Meyer A, Sorichter S, Wilkens H, Rosenkranz S, Opitz C, Leuchte H, Karger G, Speich R, Nagel C. Safety and efficacy of exercise training in various forms of pulmonary hypertension. Eur Respir J. 2012 Jul;40(1):84-92. doi: 10.1183/09031936.00123711. Epub 2012 Feb 9. PMID 22323570
- [Background] Grunig E, Maier F, Ehlken N, Fischer C, Lichtblau M, Blank N, Fiehn C, Stockl F, Prange F, Staehler G, Reichenberger F, Tiede H, Halank M, Seyfarth HJ, Wagner S, Nagel C. Exercise training in pulmonary arterial hypertension associated with connective tissue diseases. Arthritis Res Ther. 2012 Jun 18;14(3):R148. doi: 10.1186/ar3883. PMID 22709477
- [Background] Nagel C, Prange F, Guth S, Herb J, Ehlken N, Fischer C, Reichenberger F, Rosenkranz S, Seyfarth HJ, Mayer E, Halank M, Grunig E. Exercise training improves exercise capacity and quality of life in patients with inoperable or residual chronic thromboembolic pulmonary hypertension. PLoS One. 2012;7(7):e41603. doi: 10.1371/journal.pone.0041603. Epub 2012 Jul 25. PMID 22848542
- [Background] Becker-Grunig T, Klose H, Ehlken N, Lichtblau M, Nagel C, Fischer C, Gorenflo M, Tiede H, Schranz D, Hager A, Kaemmerer H, Miera O, Ulrich S, Speich R, Uiker S, Grunig E. Efficacy of exercise training in pulmonary arterial hypertension associated with congenital heart disease. Int J Cardiol. 2013 Sep 20;168(1):375-81. doi: 10.1016/j.ijcard.2012.09.036. Epub 2012 Oct 5. PMID 23041100
- [Background] Halank M, Einsle F, Lehman S, Bremer H, Ewert R, Wilkens H, Meyer FJ, Grunig E, Seyfarth HJ, Kolditz M, Wieder G, Hoffken G, Kollner V. Exercise capacity affects quality of life in patients with pulmonary hypertension. Lung. 2013 Aug;191(4):337-43. doi: 10.1007/s00408-013-9472-6. Epub 2013 May 17. PMID 23681593
- [Background] Kabitz HJ, Bremer HC, Schwoerer A, Sonntag F, Walterspacher S, Walker DJ, Ehlken N, Staehler G, Windisch W, Grunig E. The combination of exercise and respiratory training improves respiratory muscle function in pulmonary hypertension. Lung. 2014 Apr;192(2):321-8. doi: 10.1007/s00408-013-9542-9. Epub 2013 Dec 13. PMID 24338088
- [Background] Ehlken N, Lichtblau M, Klose H, Weidenhammer J, Fischer C, Nechwatal R, Uiker S, Halank M, Olsson K, Seeger W, Gall H, Rosenkranz S, Wilkens H, Mertens D, Seyfarth HJ, Opitz C, Ulrich S, Egenlauf B, Grunig E. Exercise training improves peak oxygen consumption and haemodynamics in patients with severe pulmonary arterial hypertension and inoperable chronic thrombo-embolic pulmonary hypertension: a prospective, randomized, controlled trial. Eur Heart J. 2016 Jan 1;37(1):35-44. doi: 10.1093/eurheartj/ehv337. Epub 2015 Jul 31. PMID 26231884